CLINICAL TRIAL: NCT03181802
Title: Are Paraspinous Intramuscular Injections of Botulinum Toxin A (BoNT-A) Efficient in the Treatment of Chronic Low-back Pain?
Brief Title: Are Paraspinous Intramuscular Injections of Botulinum Toxin A (BoNT-A) Efficient in the Treatment of Chronic Low-back Pain (LBP)?
Acronym: BoNT-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX2003
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This study was a randomized, double-blinded, placebo-controlled phase 3 trial comparing Intramuscular injections of botulinum toxin A to a placebo in patients with chronic low-back pain (LBP)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin A (Experimental)
  Interventions: Drug: Botox
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Botox — single injection of 200 International Unit of BoNT-A in 10 bilateral paravertebral intramuscular points for treating chronic LBP
  Arms: botulinum toxin A
Drug: Placebos — 4 ml of physiological serum injected intramuscularly into the lumbar paravertebral muscles.
  Arms: Placebo

SUMMARY:
Studying the therapeutic effect of paravertebral injections of BoNT-A (botulinum toxin A) requires further studies to confirm the reported short-term therapeutic effect and to determine potential predictive factors of efficacy.

DETAILED DESCRIPTION:
This study was a randomized, double-blinded, placebo-controlled phase 3 trial comparing BoNT-A Type A injections to a placebo in patients with chronic Low-back Pain (LBP). This superiority trial obtained support from the French Hospital Clinical Research Project (PHRC) and the approval of a French ethics committee (2003/02) ("Comité Sud-Ouest et Outre-Mer III", consent obtained in February 2003).

The number of participants included in the study was chosen to be similar as those included in previous studies, that showed a strong positive effect of BoNT-A injections on LBP. Furthermore, the design of our study (i.e. a crossover) increased the power of the statistical analysis. A scientific committee has been solicited at this step, after including 19 patients, to assess the results.

ELIGIBILITY:
Inclusion Criteria:

* LBP defined as a pain located between the thoracic lumbar hinge and the gluteal sulcus, where pain had evolved over a period of 6 months despite well conducted medical treatment, self-assessed lumbar pain intensity over 50 millimeters long on a visual analogue scale of 100 millimeters (0=no pain; 100=maximal pain),
* having been on sick leave for 60 or more days in the year preceding the inclusion (in order to include patients with high consequences of chronic low-back pain on their work),
* same long-term chronic pain treatment for at least 6 weeks

Exclusion Criteria:

* age under 18 or over 55 years (to avoid secondary causes of low back pain, like spinal tumor),
* ongoing pregnancy or breast-feeding,
* a neuromuscular pathology (myasthenia gravis, amyotrophic lateral sclerosis, myopathy, polymyositis), aminoglycoside treatment at the time of inclusion,
* skin infection at injection points,
* diabetes and alcoholism (in order to avoid other etiologies of chronic pain),
* a history of injecting BoNT-A A,
* anticoagulation treatment, sciatica,
* suspected spinal inflammatory disorder (spondylitis, inflammatory rheumatism, tumoral pathology),
* a failed back surgery syndrome (when surgery failed to relieve low-back pain), - incapacity to stand, cardiorespiratory deficiency which does not allow the isokinetic exploration of the spinal muscles,
* cognitive disorders limiting patient participation,
* conflicts of interest owing to existing pain (unconsolidated work accident, ongoing damage compensation).
* Spine infection, tumour or trauma had been specifically excluded by an MRI done by all patients before the inclusion in the present study.
* No patient was allowed to take opiates during the time of the study,
* facet joint injections were also not permitted during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-11-18 (Actual); Primary Completion 2005-05-05 (Actual); Study Completion 2005-05-08 (Actual)

PRIMARY OUTCOMES:
effect of paravertebral injections of BoNT-A, 30 days after its administration in chronic LBP sufferers. | Day 30
  Pain intensity was measured on a horizontal visual analogue scale (VAS) 100 mm long, with " no pain " written on one end and " maximum pain " on the other. The question asked was: "How was the intensity of your LBP over the last 8 days?"

SECONDARY OUTCOMES:
Evaluate the analgesic effect of paravertebral injections of BoNT-A, 90 days after its administration in chronic LBP sufferers. | Day 90
  Initial pain was detailed as follows: Immediate average LBP was recorded on VAS at the first injection
Measure the impact of paravertebral injections of 200 IU of BoNT-A in a single administration on lumbar stiffness and on spinal extensor muscle strength in patients with chronic LBP. | Day 30
  Lumbar pain intensity was measured on a horizontal visual analogue scale 100 mm long, with " no pain " written on one end and "maximum pain" on the other. The question asked was: "How was the intensity of your LBP over the last 8 days?" The question asked was: "How was the intensity of your LBP over the last 8 days?"
Measure the impact of paravertebral injections of 200 IU of BoNT-A in a single administration on lumbar stiffness and on spinal extensor muscle strength in patients with chronic LBP. | Day 120
  Lumbar pain intensity was measured on a horizontal visual analogue scale 100 mm long, with " no pain " written on one end and "maximum pain" on the other. The question asked was: "How was the intensity of your LBP over the last 8 days?" The question asked was: "How was the intensity of your LBP over the last 8 days?"

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu DE SEZE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster et al., 2001 and Machado et al., 2016
- [Derived] Cogne M, Petit H, Creuze A, Liguoro D, de Seze M. Are paraspinous intramuscular injections of botulinum toxin a (BoNT-A) efficient in the treatment of chronic low-back pain? A randomised, double-blinded crossover trial. BMC Musculoskelet Disord. 2017 Nov 15;18(1):454. doi: 10.1186/s12891-017-1816-6. PMID 29141611
- See also: Oxford Centre for Evidence-Based Medicine 2011 Levels of Evidence — http://www.cebm.net/wp-content/uploads/2014/06/CEBM-Levels-of-Evidence-2.1.pdf